CLINICAL TRIAL: NCT04542382
Title: Identification and Validation of Biomarkers for Breast Cancer Resistance Protein
Brief Title: Identification and Validation of Biomarkers for Breast Cancer Resistance Protein (BCRP)
Acronym: BCRPmarker
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20-30638
Record Dates: First submitted 2020-08-25; First posted 2020-09-09 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteers
Keywords: membrane transporter; drug-drug interaction; rosuvastatin; eltrombopag; biomarker
MeSH Terms: interventions — Rosuvastatin Calcium; eltrombopag

STUDY DESIGN:
Intervention Model Description: This is a single center, an open-label, non-randomized, fixed-sequence study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo and Rosuvastatin (Experimental): Subjects will be dosed with placebo tablet and Rosuvastatin 10mg tablet
  Interventions: Drug: Rosuvastatin
- Eltrombopag and Rosuvastatin (Experimental): Subjects will be dosed with Eltrombopag 75mg tablet and Rosuvastatin 10mg tablet
  Interventions: Drug: Rosuvastatin (Inhibitor arm); Drug: Eltrombopag

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin will be administered as follows:
  Day 1: single dose of 10 mg Rosuvastatin tablet.
  Other Names: Crestor
  Arms: Placebo and Rosuvastatin
Drug: Rosuvastatin (Inhibitor arm) — Rosuvastatin will be administered as follows:
  Day 8: single dose of 10 mg Rosuvastatin tablet.
  Other Names: Cresto
  Arms: Eltrombopag and Rosuvastatin
Drug: Eltrombopag — Eltrombopag will be administered as follows:
  Day 8: single dose of 75 mg Eltrombopag tablet.
  Other Names: Promacta
  Arms: Eltrombopag and Rosuvastatin

SUMMARY:
This is an open-label, non-randomized, fixed-sequence study. Subjects will undergo a rosuvastatin phase and eltrombopag and rosuvastatin phase to identify biomarkers for Breast Cancer Resistance Protein (BCRP).

DETAILED DESCRIPTION:
Membrane transporters are critical in the absorption, distribution and elimination of drugs, and are important target sites for drug-drug interactions (DDIs). During drug development, clinical studies characterizing transporter-mediated DDIs are frequently required. There has been enormous interest in identifying and validating serum biomarkers or surrogate probes to be used in predicting in vivo (clinical) DDIs. These biomarkers could complement in vitro studies, reducing false positive and false negative predictions, as well as the cost and time required for clinical development.

In this open-label, non-randomized, fixed-sequence study, subjects will undergo a rosuvastatin phase and eltrombopag and rosuvastatin phase to identify biomarkers for a membrane transporter known as Breast Cancer Resistance Protein (BCRP). The primary goal of this study is to validate and discover BCRP candidate biomarkers in a focused clinical DDI study with healthy volunteers to determine whether they can serve as clinical biomarkers for BCRP-mediated DDIs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as judged by medical examination, medical history and normal biochemical and hematological measures.
* Normal urinalysis and renal function
* Male subjects weighing ≥ 50 kg and female subjects weighing ≥ 45 kg.
* Understand the nature and purpose of the study and provide informed consent.

Exclusion Criteria:

* Subjects who are pregnant, breastfeeding, or unwilling to practice non-hormonal forms of birth control during participation in the study.
* Self-reported drug allergies to rosuvastatin or eltrombopag
* Subjects that have smoked cigarettes, have smoked or ingested THC/marijuana or have used illegal substances (i.e., opiates, cocaine) in the past year.
* Subjects with any disease affecting or impairing the function of the liver, kidney or heart.
* Subjects with any blood or coagulation disorders.
* Subjects with diabetes mellitus, hyperthyroidism, hypothyroidism, cardiovascular disease, glaucoma.
* Subjects with gastrointestinal disease, gastrointestinal disorder, or gastrointestinal surgery.
* Subjects with known infection with HIV, Hepatitis B (HBsAg) or Hepatitis C (no laboratory diagnostics concerning these diseases will be performed within the present study).
* Subjects that are taking prescription (i.e., birth control pills), non-prescription and dietary supplements (i.e., turmeric, quercetin, kaempferol, Gingko biloba) within seven days of receiving the study dose in each phase of the study.
* Subjects with a condition, disease, or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* Female subjects undergoing treatment for infertility or hormone replacement therapy.
* Subjects with abnormal laboratory results at screening as judged by the investigator or study physician.
* Participating in another research study while participating in this research study.
* Subjects that ingest grapefruit, grapefruit juice or grapefruit extract within seven days of receiving the study dose in each phase of the study.
* Non-English speaking.
* Subject has any signs or symptoms that are consistent with COVID-19. Per current CDC recommendations this includes subjects with the symptoms cough or shortness of breath or difficulty breathing, or at least two of the following symptoms: fever, chills, repeated shaking with chills, muscle pain, headache, sore throat or new loss of taste/smell. In addition, the subject has any other findings suggestive of COVID-19 risk in the opinion of the investigator.
* Subject tests positive for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) by a molecular diagnostic test (i.e., COVID19 RNA test) performed during the screening visit.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetics of co-administration of rosuvastatin and eltrombopag in healthy volunteers. | 24 and 72 hours
  Mean difference in area under the curve (AUC) between rosuvastatin 10mg + placebo versus rosuvastatin 10mg + eltrombopag 75mg
Composite of pharmacokinetics of co-administration of rosuvastatin and eltrombopag in healthy volunteers. | 24 hour
  Mean difference in Cmax between rosuvastatin 10mg + placebo versus rosuvastatin 10mg + eltrombopag 75mg

SECONDARY OUTCOMES:
Composite of BCRP biomarkers of co-administration of rosuvastatin and eltrombopag in healthy volunteers. | 24 and 72 hours
  Mean difference in BCRP biomarker Cmax between rosuvastatin 10mg + placebo vs rosuvastatin 10mg + eltrombopag 75mg

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Giacomini, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- Ucsf Ctsi Crc, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No